CLINICAL TRIAL: NCT04781829
Title: Use of a Rapid Diagnostic Test for Antibiotic De-escalation in Severe Community Acquired Pneumonia
Acronym: BioFire
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID pandemic precluded trial initiation. No longer clinical equipoise
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Wunderink, Professor of Medicine, Pulmonary and Critical Care, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00210610
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Intervention Model Description: Physician-specific Step Wedge
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Critically ill patients with pneumonia will be treated with an antibiotic strategy at the discretion of the treating clinician
- Interventional (Experimental): Critically ill patients with pneumonia will be treated with an antibiotic strategy based on results from the BioFire Pneumonia Panel
  Interventions: Diagnostic Test: BioFire Pneumonia Panel

INTERVENTIONS:
Diagnostic Test: BioFire Pneumonia Panel — Treatment based on an algorithm that recommends antibiotic choices based on bacteria/virus detected by BioFire Pneumonia Panel
  Arms: Interventional

SUMMARY:
The purpose of this study is to conduct an open-label step-wedge pilot clinical trial to compare an antibiotic strategy based on routine use of a novel rapid diagnostic test to usual care in critically ill adults with severe community acquired pneumonia (SCAP). We hypothesize that when results from a rapid diagnostic test (RDT) are used to guide antibiotic therapy, broad-spectrum antibiotic exposure will be reduced in critically ill patients with SCAP without an increase in adverse events.

DETAILED DESCRIPTION:
The purpose of this study is to conduct an open-label step-wedge pilot clinical trial to compare an antibiotic strategy based on routine use of a novel rapid diagnostic test to usual care in critically ill adults with severe community acquired pneumonia (SCAP). We hypothesize that when results from a rapid diagnostic test (RDT) are used to guide antibiotic therapy, broad-spectrum antibiotic exposure will be reduced in critically ill patients with SCAP without an increase in adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older with known or suspected community-acquired pneumonia who are admitted to the MICU Service
2. Meets one of the following:

   1. Have or plan to obtain a bronchoalveolar lavage (BAL)
   2. Have or plan to obtain a quantitative endotracheal aspirate sample
   3. Have already produced a high-quality sputum sample if not intubated
3. Primary MICU attending and fellow willing to base antibiotic therapy on results of RDT

Exclusion Criteria:

1. Subjects with confirmed extrapulmonary infection requiring antibiotics outside the usual treatment for SCAP, with the exception of suspected uncomplicated urinary tract infection
2. Neutropenic fever, defined as absolute neutrophil count <1000/mm3 and absence of infiltrate on available chest imaging
3. Chronic airway infection, defined as cystic fibrosis, lung transplant, or non-CF bronchiectasis
4. Patient/surrogate refusal
5. Inability to perform BAL, NBBAL, quantitative ETA, or produce a high-quality sputum sample prior to 48 hours from hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-15 (Estimated); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
Narrow-spectrum Antibiotic Treatment | 14 days
  A quantitative tool that reflects how broad or narrow antibiotic is

IPD SHARING:
Plan to Share IPD: No